CLINICAL TRIAL: NCT00972127
Title: Changes in the Renal Excretion of Neramexane by Acidification of Urinary pH Open-Label, Randomized, Single Center, Multiple Dose, 2-Period, 2-Sequence, Crossover Study With and Without Application of a Urinary pH Acidification Regimen
Brief Title: Changes in the Renal Excretion of Neramexane by Acidification of Urinary pH Study With and Without Application of a Urinary pH Acidification Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Dr. med. Horst Jürgen Heuer, AAIPharma Deutschland GmbH & Co. KG
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 92579/TI/1004
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
MeSH Terms: interventions — neramexane

INTERVENTIONS:
Drug: Neramexane — 25 mg or 2x25mg tablets

SUMMARY:
Primary:

* To assess the influence of acidified urinary pH on the renal excretion of Neramexane

Secondary:

* To assess the influence of acidified urinary pH on the renal excretion of N-OH Neramexane
* To assess the steady state plasma pharmacokinetics (PK) of Neramexane and N-OH Neramexane under physiological conditions and under the conditions of urine acidification
* To assess safety and tolerability of a repeated dose treatment of Neramexane under physiological conditions and under the conditions of urine acidification

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subject of any ethnic origin, who is able to read, to write and fully understand German language
* Aged 18 to 45 years
* BMI of 18-28 kg/m2 and a body weight of 50-90 kg
* Willing and able to provide written informed consent after having been informed of the requirements and the restrictions of the study
* Female subject of childbearing potential must agree to use an effective method of birth control such as sexual abstinence, vasectomised partner, non hormonal IUDs or double contraception methods (e.g., condom with spermicide cream)

Exclusion Criteria:

* History of clinically relevant allergy or known hypersensitivity to Neramexane/Memantine/Amantadine and their derivatives
* History of clinically relevant allergy or known hypersensitivity to Ammonium Chloride
* Exposure to another investigational agent within the last two months before Day 1 of Period 1
* History of clinically relevant allergy or known hypersensitivity to any inactive ingredient in any of the used investigational products or tool substances
* Lactating or pregnant female or female planning to become pregnant during study conduct or within 2 months after end of study. Male planning to beget children during study conduct or within 2 months after end of study
* Any contraindications which are indicated in the topically valid SPC for Extin®N: acidosis, gastritis, gastro-intestinal ulcer, hepatic or renal insufficiency, hypokalemia

Lack of suitability for the trial

* Any evidence of a significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, endocrinological, metabolic (acidosis), psychiatric or other disease at screening
* History of malignancy
* Any clinically relevant deviation in clinical or laboratory assessment
* Clinically relevant abnormalities in the 12-lead ECG which in the discretion of the investigator and the Merz scientific expert might affect the study objectives
* Systolic blood pressure <95 mmHg or >150 mmHg or diastolic blood pressure < 50 mmHg or >90 mmHg in supine position
* Pulse rate <45 or >100 beats per minute
* Clinically relevant chronic or acute infections
* Acute or chronic disease, especially psychiatric or neurologic disorders
* Current evidence of hypokalemia (= below lower limit of laboratory normal range plus 0.3 mmol/l as safety margin)
* History of alcohol or drug dependence within the last 2 years
* Alcohol consumption averaging more than 40 g for male and more than 20 g for female subject daily within the last year
* Regular caffeine consumption averaging more than 1 L of coffee and/or tea daily or more than 1 L of caffeine-containing lemonades per day within the last year
* Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal products (e.g. acute inflammations, gastrointestinal disease, cholecystectomy, resection of small or large intestine, etc.)
* Use of any prescribed medication for four weeks prior to the first administration of IMP.

  * Regular use of over-the-counter [OTC] drugs in the 4 weeks prior to the first administration of the IMP
  * Occasional use of OTC drugs (except paracetamol, maximum 1 g/day) within the 2 weeks prior to the first administration of the IMP
  * Stable intake of thyroid hormone substitution will be allowed.
* Use of any food, food supplement or medication known to induce or inhibit CYP3A4 or other cytochrome P450 enzymes within two weeks preceding the start of the study (Day 1), e.g. grapefruit, St. John's wort
* Special diet, e.g. vegetarian
* Female subject who employed any form of hormonal contraception within 2 months prior to Day 1 (e.g. oral contraceptives, hormone releasing intrauterine contraceptive devices [IUDs], etc.)
* Consume of xanthine derivates (including caffeine) within two days prior to Day 1
* Smoker and user of snuff, nicotine replacement and chewing tobacco
* Previous enrolment into the clinical phase of the current study
* Positive results in any of the serology tests
* Blood donation of more than 450 mL within 60 days prior to Day 1
* Positive pregnancy test, if female
* Positive drug screen or alcohol test

Administrative reasons

* Lack of willingness or inability to co-operate adequately
* Employee or direct relative of an employee of the CRO or Merz Pharmaceuticals GmbH
* Lack of ability or willingness to give informed consent
* Vulnerable subject (e.g. person kept in detention)
* Anticipated non-availability for study visits/procedures
* Inability to follow study procedures and investigator instructions adequately

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)